CLINICAL TRIAL: NCT03916939
Title: Contribution of Osteopathic Treatment to Alcohol Withdrawal Syndrome in Hospitalized Adult Patients
Brief Title: Osteopathic Treatment to Alcohol Withdrawal Syndrome
Acronym: OSTEOOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Ecole Supérieur d'Ostéopathie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OSTEOOL
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2022-06

CONDITIONS: Alcohol Withdrawal
MeSH Terms: interventions — Osteopathic Physicians

STUDY DESIGN:
Who Masked: Participant
Masking Description: simulated osteopathy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathy (Experimental): osteopathic treatment
  Interventions: Other: osteopathy
- simulated osteopathy (Placebo Comparator): simulated osteopathic treatment
  Interventions: Other: simulated osteopathy

INTERVENTIONS:
Other: osteopathy — osteopathy treatment
  Arms: Osteopathy
Other: simulated osteopathy — simulated osteopathic sessions
  Arms: simulated osteopathy

SUMMARY:
The alcohol withdrawal syndrome has a hierarchical symptomatology depending on the severity (minor, moderate or severe). These signs express a state of psychic, behavioral and physical deprivation.

The management of withdrawal syndrome involves the establishment of pharmacological and psychosocial interventions.

Osteopathy is an exclusively manual practice whose purpose is to overcome the dysfunction of mobility of tissues of the human body. It can be used as a complementary treatment when a specific support is put in place. The purpose of this study is to examine the effectiveness of osteopathy in reducing alcohol withdrawal symptoms in adult patients.

DETAILED DESCRIPTION:
The use of osteopathic techniques for facial equilibration decreases the severity of withdrawal symptoms experienced by patients hospitalized in a weekday hospital.

ELIGIBILITY:
Inclusion Criteria :

* Age> 18 years
* Patient hospitalized for a programmed alcohol withdrawal
* Patient not abstinent with alcohol before hospitalization
* Signed informed consent

Exclusion Criteria :

* Minor patient
* Patient with an addiction other than alcohol (except tobacco and benzodiazepines)
* Previous participation in the OSTEOOL study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2023-12-13 (Estimated); Study Completion 2024-02-13 (Estimated)

PRIMARY OUTCOMES:
Cushman score (0 to 27) | Day one
  comparison between the two groupe of the cushamn socre between 11:30 am and 00:00 pm. questionary for alcohol dependency

SECONDARY OUTCOMES:
CIWA Ar (Clinicial Institute Withdrawal Assessment - Alcohol Revised) test (0 to 67) | day 0
  comparison between the two groups with this questionary for alcohol withdrawal
CIWA Ar test (0 to 67) | day 1
  comparison between the two groupe with this questionary for alcohol withdrawal
CIWA Ar test (0 to 67) | day 2
  compariason between the two groups with this questionary for alcohol withdrawal
CIWA Ar test (0 to 67) | day 3
  comparison between the two groups with this questionary for alcohol withdrawal
CIWA Ar test (0 to 67) | day 4
  comparison between the two groups with this questionary for alcohol withdrawal
cardiac frequency (beat per minute) | day 1
  mesurement of cardiac frequency and compaaison between the two groups
cardiac frequency (beat per minute) | day 3
  mesurement of cardiac frequency and comparison between the two groups
cardiac frequency (beat per minute) | day 4
  measurement of cardiac frequency and comparison between the two groups
quality sleep scale (0 to 5) | day 0
  comparison between the two groups with sleep score
quality sleep scale (0 to 5) | day 1
  comparison between the two groups with sleep score
quality sleep scale (0 to 5) | day 2
  comparison between the two groups with sleep score
quality sleep scale (0 to 5) | day 3
  comparison between the two groups with sleep score
quality sleep scale (0 to 5) | day 4
  comparison between the two groups with sleep score
quantity of benzodiazepine mg per 24 hours | day 2
  comparison between the two groups of benzodiazepin use
quantity of benzodiazepine (mg per 24 hours) | day 3
  comparison between the two groups of benzodiazepin use
quantity of benzodiazepine (mg per 24 hours) | day 4
  comparison betwenn the two groups of benzodiazepin use
Cushmamn score (0 to 27) | day 3
  comparison between the two groups of the Cushamn score between 11:30 am and 00:00 pm

CONTACTS AND LOCATIONS:
Locations (1):
- Chi Creteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No